CLINICAL TRIAL: NCT06121739
Title: Participatory Design and Feasibility of a Multicomponent Intervention to Improve the Well-being of Elementary School Children After the COVID-19 Pandemic
Brief Title: Child and Adolescent Mental Health Literacy for Primary Schools Teachers. A Multicomponent Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FONIS SA21I0143
Record Dates: First submitted 2023-09-22; First posted 2023-11-08 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2023-05

CONDITIONS: Child Mental Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child Mental health Literacy Program (Experimental): Teachers from four schools will attend a nine-session workshop on mental health literacy. They will participate in face-to-face sessions and use an online platform.
  Interventions: Behavioral: Child Mental Health Literacy Program
- Control (No Intervention): Teachers from four schools will not receive any additional mental health training

INTERVENTIONS:
Behavioral: Child Mental Health Literacy Program — The workshop has a participant-oriented character, seeking to apply the more theoretical contents to the local school context. It has four units and a total of nine modules, each lasting 90 or 120 minutes, with reference material on an educational platform. The topics are : 1) the person behind the role of educator; 2) the school community and its influence on the healthy development of students; 3) the expected development and its alterations in the different evolutionary stages; 4) common and differential factors of child and adolescent mental health disorders; 5) Stigma in Mental Health; 6) screening, the first care, and use of devices for the prevention and treatment of mental health disorders in children and adolescents.
  Arms: Child Mental health Literacy Program

SUMMARY:
Child mental health (CMH) is crucial for lifelong well-being. Early prevention and intervention are vital for public health, yet Chile faces a high prevalence of CMH issues, particularly in children aged 4 to 11. Schools play a key role in addressing these problems, but there's a lack of coordination within the systems (Schools and Health Centers). This project aims to enhance children's mental health and the school community through a biopsychosocial approach, emphasizing social support.

The intervention consists of two parts:

1. Developing an online CMH literacy program for primary school teachers in Public Educational Establishments (EEPs). It's designed through collaboration with stakeholders, focusing on the specific needs of participating schools.
2. Enhancing the coordination of the CMH network in Valparaíso, involving community, health, and education stakeholders in two neighborhoods. This will be done by using "ECO Barrio Solidario" program and aligning it with local health initiatives.

The project spans two years and focuses on four EEPs in Valparaíso. In the first year, the literacy intervention is constructed in partnership with each school, including program objectives, methodology, and scope. An online platform with educational videos will be created. The "ECO-Barrio Network" will connect with local agencies involved in child MH. In the second year, the intervention will be implemented in four of the eight recruited schools, while the other four serve as a control group. Subsequently, the remaining four schools will receive the intervention. Evaluation will consider acceptability, feasibility, and effectiveness, assessing faculty CMH knowledge, timely research, and reduced wait times for healthcare and child protection services.

DETAILED DESCRIPTION:
This proposal aims to build "school communities" based on Public Schools (PS), with the goal of promoting children's mental health (MH) and detecting early MH issues in students, providing them with initial support and coordinated referrals for treatment.

To achieve this, a participatory multicomponent intervention is proposed to promote the MH of children attending basic education. The components of this grant are: 1) a Child Mental Health (CMH) Literacy program for PS teachers, which will be constructed in a participatory manner with them and other key stakeholders; and 2) the coordination of the local network of child and adolescent mental health care, including various levels of complexity (community, primary care, and specialized care). This network is based on the ECO-BARRIO SOLIDARIO strategy with adaptations according to the new socio-sanitary context.

Given the nature of a pilot project that seeks to evaluate the feasibility of this intervention initially, it is proposed to implement it in two neighborhoods of Valparaíso, with a random selection of 8 PS with primary education in each of these neighborhoods. After the program's implementation, the initial effectiveness of the CMH literacy component will be evaluated with the teachers.

The process of participatory construction of the CMH Literacy program will be developed during the first 12 months of the project. It will involve working with representatives of the academic staff of these EPs (teachers, para-teachers, directors, and others), parents, students, directors of the Local Education Service (SLEP) of Valparaíso, and representatives of the ECO-Barrio network.

Through working groups and individual interviews with key stakeholders, a survey of objectives, methodology, and contents of the CMH Literacy program will be conducted. Due to the health situation resulting from the COVID-19 Pandemic and the current development of Information and Communication Technologies (ICTs), an asynchronous and synchronous online program is proposed. This program will be based on recorded video educational capsules and discussion groups with CMH specialists, respectively. There will be an evaluation at the beginning and at the end of the course to measure acquired knowledge and the level of satisfaction with the methodology and content, among other factors. The course will be free and certified by the Faculty of Medicine of the University of Valparaíso. Certification will be automatic for those who fulfill all the requirements on the online platform, which will be accessible from computers or mobile phones. The total duration of the course should be between 3 to 4 months.

Parallel to the construction of the CMH Literacy program for teachers, the "ECO BARRIO SOLIDARIO" strategy will be implemented in one of the neighborhoods with modifications according to the new health and contextual scenario. This strategy will be called the "ECO-Barrio Network." The ECO-Barrio Network strategy is feasible to replicate since there are Joint Health-Education Commissions (COMSE) in Primary Health Care (PHC) aiming to connect CESFAM with the Educational Establishments that converge in a territory to develop strategies for prevention, participation, and health promotion in educational communities. Particularly in Valparaíso, since 2020 and in response to the socio-health crisis due to COVID-19, a COMSE 2.0 strategy has been developed. Its objectives include reactivating COMSE meetings with the participation of Mental Health Managers from each school, the psychosocial duo of the PHC health team, and the participation and promotion officer of CESFAM. It also aims to develop a socio-educational process for COMSE participants to improve the referral and follow-up of cases from the educational community to PHC, as well as the development of prevention and promotion strategies in MH. Additionally, it intends to create a containment, prevention, and promotion device in MH for the educational communities of the educational establishments associated with each CESFAM. These new objectives of COMSE 2.0 align with the ECO-Barrio Network strategy and this project.

The contribution of the ECO-Barrio Network strategy will be to systematically convene potential participants of COMSE, including all relevant participants in the CMH of that neighborhood (Health from primary care with the CESFAM and CECOF that correspond, plus specialized care with the Outpatient Unit of Child and Adolescent Psychiatry of the Psychiatric Hospital of Salvador (HDS), SENAME in its different programs, and others such as Life Skills (HPV)). In addition, through articulation with the Secondary level of Mental Health and the link with the Chair of Child Psychiatry at the University of Valparaíso, the ECO-neighborhood Network will be able to organize and provide training, generate a case monitoring system on an online platform, and evaluate the implementation process in the two selected neighborhoods, which will serve as input for potential replication in other territories of Valparaíso.

This project promotes and strengthens the co-construction of responses and articulated strategies for children, highlighting the community's role as the central axis of action. This multimodal intervention can help address the significant increase in CMH problems resulting from the COVID-19 pandemic and the social crisis. It is also considered a useful model for stable implementation throughout Chile since it includes interventions to increase knowledge and problem-solving skills in CMH for faculty, a component not addressed in other research or management instances known in our country.

The relevance and feasibility of scaling up to the rest of the country are ensured through the participatory process involving local key stakeholders, as well as the participation of SLEP, Health, and the Municipality of Valparaíso. This proposal aligns with the community approach outlined in the National Plan for MH and Psychiatry 2017-2025 and aims to respond to the increase in MH problems in the child-adolescent population and reduce social inequalities that persist in our country despite macroeconomic growth.

RESEARCH QUESTION Is a multi-component intervention, constructed in a participatory manner and with a territorial perspective, feasible and effective in improving the mental health of children in public educational establishments, identifying, and treating those in need? RESEARCH HYPOTHESES OR ASSUMPTIONS

1. Teachers who participate in a Child Mental Health Literacy program can significantly improve their knowledge regarding the identification of these problems and the delivery of initial aid.
2. The establishments that participate in this training program can significantly improve the detection rate of children with mental health problems.
3. The relevance of the diagnosis made by teachers when referring children with mental health problems to the corresponding CESFAM is greater than 80%.
4. The health-education networks where an intervention is carried out to articulate the referral of girls and boys with mental health problems can reduce the waiting time between referral and the first health care.

OBJECTIVES GENERAL OBJECTIVE Evaluate the effectiveness and feasibility of a multicomponent intervention, constructed in a participatory manner and with a territorial approach, to improve the mental health of children in public educational establishments, identifying and treating those in need in a timely manner.

SPECIFIC OBJECTIVES

1. Design the contents of a Child Mental Health (CMH) Literacy program with teachers of Public Educational Establishments (PS) and key actors from the commune of Valparaíso in a participatory manner.
2. Implement the strategy of articulation in a network of CMH (ECO-Neighborhood Network) between schools, Primary and Secondary Health Care, Municipality, collaborating agencies of SENAME, and other relevant programs in two territories of the commune of Valparaíso.
3. Evaluate whether the children of PS that are part of the strategy of the ECO-Neighborhood Network have better levels of mental health than those who do not participate in this network.
4. Evaluate the impact of the CMH Literacy program for teachers on knowledge acquisition and the level of satisfaction with the methodology and content.
5. Evaluate the impact of the ECO-Neighborhood Network strategy on the reduction of waiting times between referral and first care for children in PHC and specialized care.
6. Determine the diagnostic relevance of the cases referred by teachers to PHC. METHODOLOGY This research will use a mixed-methods approach, combining quantitative and qualitative methods to evaluate the effectiveness and feasibility of the intervention.

Quantitative Component:

* Pre- and post-test evaluations will be conducted to measure the impact of the CMH Literacy program for teachers on their knowledge acquisition and the level of satisfaction with the program.
* Comparison of mental health outcomes in children from PS participating in the ECO-Neighborhood Network with those who do not participate.
* Analysis of waiting times between referral and first care for children in PHC and specialized care in the ECO-Neighborhood Network compared to those not participating.

Qualitative Component:

* In-depth interviews with key stakeholders, including teachers, parents, students, and health professionals, to gather insights into the feasibility and acceptability of the intervention.
* Focus group discussions to explore the experiences and perceptions of participants in the CMH Literacy program.
* Process evaluation of the implementation of the ECO-Neighborhood Network.

ELIGIBILITY:
Inclusion Criteria:

* All the teachers in the participating schools
* Both gender

Exclusion Criteria:

* Lack of informed consent.
* Teachers who are leaving or not planning to be in the school at any time during 2023

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Teachers' level of knowledge about infant mental health | Immediately prior to the intervention and after the completion of the intervention up to 4 weeks
  Teachers' level of knowledge, using the "Children's Mental Health Questionnaire for Educators," scores range from 0 to 13, with higher scores indicating better knowledge of mental health.
Feasibility of the intervention assessed by the proportion of teachers who complete the workshop | Immediately after the completion of the intervention up to 4 weeks
  Level of retention of teachers in the intervention will be estimated through the proportion of teachers who complete the course of all those who started it.
Satisfaction assessed by a Likert Survey | Immediately at the conclusion of each session
  Level of satisfaction of teachers with the intervention, an ad hoc survey will be used, with Likert questions for each module of the training course
Rate of accuracy for referral of children | Between 8 to 16 weeks after the completion of the intervention
  with suspected psychiatric disorders from the school to health care. Each "case" referral will apply the Strength and Difficulties Questionnaire (SDQ). 25 items (scale 0-2)

SECONDARY OUTCOMES:
Rates of referral of mental health problems in children | Through study completion, an average of 10 months
  Rates of referral of mental health problems in children from the school to primary health center,
Waiting time between referral to first attention in the health center | Through study completion, an average of 12 months
  Waiting time between referral from the educational establishment to professional care at the corresponding CESFAM
Level of interest of teachers in the intervention | At the beginning of the intervention, for up to 4 weeks
  It is estimated through the percentage of teachers who agree to start the training course, out of the total number of teachers who were invited

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio Local de Educación (SLEP), Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocol (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT06121739/Prot_SAP_ICF_000.pdf
  • Informed Consent Form: Informed Consent Form in English (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT06121739/ICF_001.pdf